CLINICAL TRIAL: NCT05755243
Title: Human Subcutaneous infLammatory Response to Glucose Sensors: Impact on the Quality of the Measure
Brief Title: Human Subcutaneous Inflammatory Response to Glucose Sensors
Acronym: TISSUESENSOR
Status: Completed | Type: Observational
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Mercedes Rigla, Director of Department, Corporacion Parc Tauli
Other Study IDs: PI18/01118
Record Dates: First submitted 2023-02-23; First posted 2023-03-06 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Inflammatory Response to Glucose Sensors
Keywords: Enzymatic glucose sensors, foreign body response

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — S.c. tissue biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Biopsy performed: after 10 days of use, the sensor is removed and the biopsy performed
  Interventions: Device: glucose sensor

INTERVENTIONS:
Device: glucose sensor — skin biopsy (punch)

SUMMARY:
The aim of the study is to describe the inflammatory response to enzimatic glucose sensors after 10 days of use and to evaluate the relationship between the magnitude of the FBR (foreign body response) with the accuracy of the sensor (MARD)

DETAILED DESCRIPTION:
Eighteen Type 1 DM patients are going to be included. Primary Objectives

1. To define the intra-individual and inter-individual variability of the macrophage count around the sensor
2. To assess whether there is a relationship between the number of macrophages, fibrosis and MARD of the MCG registry.

Secondary Objectives

To describe the histology of tissue response. This description will include:

1. HE stain: cell types, arrangement, vascular structures, signs of hemorrhage-clot. Giemsa stain: mast cells. Masson's trichrome stain: str. vascular.
2. Immunohistochemistry: Vascular assessment, characterization of macrophages

Each patient will have 1 glucose sensor inserted in the non-dominant arm. During the useful life of the sensor (10), a minimum of 4 capillary blood glucose determinations/day will be performed The sensor has a length of 8 mm and a diameter of 0.4 mm. All the necessary material will be provided, including a control diary to help the patient remember to carry out the self-control and set its time distribution.

On the last day of sensor use, it will be removed and a 4-mm punch skin biopsy will be performed 5 minutes later.

Tissue samples will be fixed in 4% formaldehyde solution, paraffin blocks made and sectioned. The resulting samples will be stained Semiquantitative determination of lymphocytes, neutrophils, mast cells, macrophages will be performed; fibrin, fibrosis, vascular proliferation and karyorrhexis

In all cases, a quantitative immunohistochemical study will be performed with x40 field counting with photographs and grid (Dako omnis with envision system) for:

Macrophages

The monitor-glucometer will be recovered for download and study of the record. The interstitial glucose - blood pairs will be made with those recorded but not used for callibration.

Glucose sensor values and insulin doses will be recover from tha medical application

ELIGIBILITY:
Inclusion Criteria:

* 1. Type 1 diabetes of more than 6 months duration, confirmed by positivity for Ab antiGAD 65 2. Be a regular user of a continuous glucose monitoring system 2. To Understand the proposed protocol and acceptance of participation.

Exclusion Criteria:

* Treatment with drugs that could potentially modify the inflammatory response during the 10 days prior to surgery (non-steroidal anti-inflammatory drugs or corticosteroids, antioxidants or platelet antiaggregants).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eighteen people diagnosed with type 1 diabetes and treated with closed-loop systems
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2022-06-21 (Actual); Primary Completion 2023-07-12 (Actual); Study Completion 2023-09-20 (Actual)

PRIMARY OUTCOMES:
Number of Macrophages sourronding the sensor | 10 days
MARD (CGM record for 10 days) | 10 days
  median absolute relative difference (BG- Sensor glucose)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Parc Tauli, Sabadell, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rigla M, Pons B, Rebasa P, Luna A, Pozo FJ, Caixas A, Villaplana M, Subias D, Bella MR, Combalia N. Human Subcutaneous Tissue Response to Glucose Sensors: Macrophages Accumulation Impact on Sensor Accuracy. Diabetes Technol Ther. 2018 Apr;20(4):296-302. doi: 10.1089/dia.2017.0321. Epub 2018 Feb 22. PMID 29470128